CLINICAL TRIAL: NCT01513174
Title: Multicenter, Randomized, Phase Ib/IIb Study to Evaluate the Efficacy and Tolerability of Gefitinib in Combination With Olaparib (AZD2281) Versus Gefitinib Alone, in Patients With EGFR Mutation Positive Advanced Non-small-cell Lung Cancer
Brief Title: Study With Gefitinib in Combination With Olaparib (AZD2281) Versus Gefitinib Alone
Acronym: GOAL
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Spanish Lung Cancer Group (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GECP10-03_GOAL; 2010-024178-21 (EudraCT Number)
Record Dates: First submitted 2011-12-11; First posted 2012-01-20 (Estimated); Results first posted 2024-06-28 (Actual); Last update posted 2024-06-28 (Actual); Status verified 2024-01

CONDITIONS: Non Small Cell Lung Cancer
Keywords: GOAL; Lung; Non small cell lung cancer; EGFR mutations
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Gefitinib; olaparib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Control Gefitinib (Active Comparator): Gefitinib will be administered once daily, continuously, in 28-day cycles, as a fixed dose of 250 mg/day.
  Interventions: Drug: Gefitinib
- Experimental: Gefitinib in combination with olaparib (Experimental): Gefitinib 250 mg once a day, in combination with olaparib (at the recommended dose in the previous Phase I study) twice a day, continuously, in 28-day cycles.
  Interventions: Drug: Gefitinib; Drug: Olaparib

INTERVENTIONS:
Drug: Gefitinib — Gefitinib 250 mg once a day, continuously, in 28-day cycles, until progression
  Other Names: Iressa
Drug: Olaparib — Gefitinib 250 mg once a day, in combination with olaparib (at the recommended dose in the previous Phase Ib study) twice a day, continuously, in 28-day cycles.
  Other Names: Lynparza
  Arms: Experimental: Gefitinib in combination with olaparib

SUMMARY:
This is a study of gefitinib plus olaparib gefitinib in combination with olaparib (AZD2281) versus gefitinib alone, in patients with Epidermal Growth Factor Receptor (EGFR) mutation positive advanced non-small-cell lung cancer.

DETAILED DESCRIPTION:
GOAL is a multicenter, randomized phase IB/II study performed in two countries, Spain and Mexico. Eligible patients were 18 years or older, treatment-naïve, pathologically confirmed stage IV NSCLC, with centrally confirmed EGFR mutations and measurable disease. Patients were randomly allocated (1:1) to receive gefitinib 250 mg daily or gefitinib 250 mg daily plus olaparib 200 mg three times daily in 28-day cycles. The primary endpoint was PFS. Secondary endpoints included overall survival (OS), response rate, safety and tolerability.

ELIGIBILITY:
Inclusion Criteria:

1. Patients age 18 years or more.
2. Histologically confirmed diagnosis of non-small-cell lung carcinoma.
3. Stage IV disease, following the Seventh Edition of the American Joint Committee on Cancer (AJCC) Cancer Staging Manual (27).
4. Tumor tissue available (according to the criterion of the specimen-processing laboratory) for EGFR mutation assessment: to be included in the study patients should present at least one EGFR mutation (exon 19 deletion or L858R with or without T790M).
5. Evidence of measurable disease per Response Evaluation Criteria in Solid Tumors (RECIST) criteria version 1.1.
6. ECOG score ≤ 2.
7. Life expectancy of ≥ 3 months.
8. For the Phase II part of the study, patients should not have received previous treatment with chemotherapy or other agents for advanced disease: chemotherapy is allowed if the initial diagnosis of the patient is limited disease and the patient has received adjuvant or neoadjuvant treatment, as long as a minimum of 6 months has passed since the end of the adjuvant and/or neo-adjuvant chemotherapy. This criterion is not mandatory to patients to be included in the Phase I part of the study (these patients are allowed to have received a prior line of treatment for advanced disease).
9. Patients with the following hematologic values:

   * Absolute Neutrophil Count (ANC) ≥1.5 x 109/L
   * Hemoglobin (Hb) ≥ 10 g/dl
   * Platelets ≥ 100 x 109/L
10. Patients with the following biochemical values:

    * Bilirubin ≤ 1.5 mg/dL
    * Aspartate aminotransferase (AST) and Alanine transaminase (ALT) < 1.5 upper limit of normality
    * Creatinine clearance ≥ 60 ml/min.
11. Patients of childbearing age of either sex must use effective contraceptive methods(barrier methods plus other birth control methods) before entering the study and while participating in the study.
12. Patients should sign an informed consent form before inclusion in the study that specifies that the clinical trial treatment entails consent for the analysis of biological samples of tumor and blood.
13. Patients must be available for clinical follow-up.

Exclusion Criteria:

1. Patients diagnosed of another neoplasm, with the exception of cervical carcinoma insitu, treated squamous cell carcinoma or superficial bladder tumor (Ta and TIS), or other malignant tumors that have received curative treatment within the last 5 years before inclusion in the study.
2. Simultaneous participation in any other study involving an investigational medicinal product, or having participated in a study less than 28 days prior to the start of study treatment.
3. Patients with HIV infection, HCV infection, coronary disease or uncontrolled arrhythmia, uncontrolled cerebrovascular disease and other clinical conditions that, in the judgment of the investigator, contraindicate the patient's participation in the study.
4. Past medical history of interstitial lung disease (ILD), drug-induced interstitial disease, radiation pneumonitis which required steroid treatment or any evidence of clinically active interstitial lung disease.
5. Pre-existing idiopathic pulmonary fibrosis evidenced by CT scan at baseline.
6. Uncontrolled seizures.
7. Patients considered requiring radiotherapy to the lung at the time of study entry or in the near future.
8. Known or suspected brain metastases or spinal cord compression, unless treated with surgery and/or radiation and stable without steroid treatment for at least 4 weeks prior to the first dose of study medication.
9. Patients unable to swallow orally administered medication and patients with gastrointestinal disorders likely to interfere with absorption of the study medication.
10. Patients who are pregnant or breastfeeding. Women of childbearing potential must have a negative pregnancy test performed within 7 days before the onset of treatment(Appendix 8).
11. Patients receiving the following classes of inhibitors of CYP3A4 (see Appendix 5 for guidelines and wash out periods):

    * Azole antifungals
    * Macrolide antibiotics
    * Protease inhibitors
12. Concomitant use of known CYP3A4 inducers such as phenytoin, carbamazepine, rifampicin, barbiturates, or St John's Wort.
13. Major surgery within 2 weeks of starting study treatment; patients must have recovered from any effects of any major surgery.
14. Significant weight loss (= 10% of body weight) in the 6 weeks before inclusion in the study.
15. Any condition that is unstable or could endanger the patient's safety and/or the patient's compliance with the study.
16. Substance abuse or clinical, psychological or social conditions that can undermine the validity of the informed consent or protocol compliance.
17. Patients who present any contraindication or suspected allergy to the products under investigation in the study. Tablets of gefitinib contain lactose: patients with rare hereditary problems of galactose intolerance, the Lapp lactose deficiency or glucose and galactose malabsorption, will not be included in this trial.
18. Contraindication for steroid use.
19. Impossibility to comply with treatment due to cultural or geographic circumstances.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 186 (Actual)
Dates: Start 2011-08 (Actual); Primary Completion 2016-07 (Actual); Study Completion 2016-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Maria Rosario García Campelo, MD, Study Chair — Hospital Teresa Herrera
Locations (5):
- Spain (5):
  - H. Germans Trias i Pujol, Badalona, Barcelona
  - ICO Hospitalet, L'Hospitalet de Llobregat, Barcelona
  - H. Teresa Herrera, A Coruña
  - H. Gen. Universitario de Alicante, Alicante
  - H. Vall d'Hebrón, Barcelona

REFERENCES:
- [Result] Garcia-Campelo R, Arrieta O, Massuti B, Rodriguez-Abreu D, Granados ALO, Majem M, Vicente D, Lianes P, Bosch-Barrera J, Insa A, Domine M, Reguart N, Guirado M, Sala MA, Vazquez-Estevez S, Caro RB, Drozdowskyj A, Verdu A, Karachaliou N, Molina-Vila MA, Rosell R; Spanish Lung Cancer Group (SLCG). Combination of gefitinib and olaparib versus gefitinib alone in EGFR mutant non-small-cell lung cancer (NSCLC): A multicenter, randomized phase II study (GOAL). Lung Cancer. 2020 Dec;150:62-69. doi: 10.1016/j.lungcan.2020.09.018. Epub 2020 Oct 3. PMID 33070053
- See also: Spanish Lung Cancer Group website — http://www.gecp.org

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Control Gefitinib | Experimental: Gefitinib in Combination With Olaparib
Started | 94 | 92
Completed | 90 | 84
Not Completed | 4 | 8
Not completed — Inclusion Error | 1 | 7
Not completed — Not receive study treatment | 3 | 1

BASELINE CHARACTERISTICS:
Population: The mITT population is defined as the set of patients included in the study who received at least one dose of the study drug. There are 182 patients in the mITT population.
Groups:
- Total: Total of all reporting groups
Arm/Group | Control Gefitinib | Experimental: Gefitinib in Combination With Olaparib | Total
Number analyzed (Participants) | 91 | 91 | 182
Age, Continuous [Mean (Standard Deviation); unit: years] | 65.97 (11.29) | 63.40 (11.39) | 65.95 (11.29)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 57 | 66 | 123
  Male | 34 | 25 | 59
Region of Enrollment [Number; unit: participants]
  Spain | 81 | 78 | 159
  Mexico | 10 | 13 | 23
Smoking status [Number; unit: participants]
  Smoker | 4 | 10 | 14
  Former smoker | 27 | 26 | 53
  Never smoker | 60 | 55 | 115
ECOG Performance Status Scale [Number; unit: participants] — ECOG Performance Status Scale: It describes a patient's level of functioning in terms of their ability to care for themself, daily activity, and physical ability
  GRADES:
  ECOG 0: Fully active. ECOG 1: Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature ECOG 2: Ambulatory and capable of all selfcare but unable to carry out any work activities; up and about more than 50% of waking hours ECOG 3: Capable of only limited selfcare; confined to bed or chair more than 50% of waking hours ECOG 4: Completely disabled ECOG 5: Dead
  participants
    ECOG 0 | 25 | 24 | 49
    ECOG 1 | 59 | 59 | 118
    ECOG 2 | 7 | 8 | 15
Bone metastasis [Number; unit: participants]
  Yes | 25 | 30 | 55
  No | 66 | 61 | 127
CNS metastasis [Number; unit: participants]
  Yes | 11 | 10 | 21
  No | 80 | 81 | 161
EGFR mutation [Number; unit: participants]
  EGFR exon 18 | 3 | 3 | 6
  EGFR exon 20 | 1 | 2 | 3
  Exon 21 L858R | 35 | 25 | 60
  del 19 | 52 | 57 | 109
  UK | 0 | 4 | 4

OUTCOME MEASURES:

1. Primary Outcome: Progression-free Survival (PFS)
Description: Defined as the length of time from the date of randomization to the date of the first documented progression of disease. "Progression is defined using Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0), as a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions"
Time Frame: From the date of randomization until end of follow up, up to 30 months.
Population: The PFS analysis is performed on the PP population
Measure: Median (Full Range); unit: Month
Arm/Group | Control Gefitinib | Experimental: Gefitinib in Combination With Olaparib
Number analyzed (Participants) | 90 | 84
Month | 10.9 [9.3 to 13.3] | 10.9 [8.6 to 13.4]
Statistical Analysis 1: Comparison: Control Gefitinib vs Experimental: Gefitinib in Combination With Olaparib; Test type: Superiority; p = 0.124, Log Rank; Hazard Ratio (HR) = 1.38, 95% CI 2-sided [1.00 to 1.92]; The initial hypothesis estimated that the median PFS for the gefitinib group would be 10 months, while the median PFS for the gefitinib/olaparib group would be 16 months, which implied a hazard ratio (HR) of 1.6

2. Secondary Outcome: Overall Survival
Description: Defined as the length of time from either the date of diagnosis or the start of the treatment that patients diagnosed with the disease are still alive.
Time Frame: From the date of randomization until end of follow up, up to 30 months
Population: The OS analysis is performed on the mITT population.
Measure: Median (Full Range); unit: Month
Arm/Group | Control Gefitinib | Experimental: Gefitinib in Combination With Olaparib
Number analyzed (Participants) | 91 | 91
Month | 23.1 [19.1 to 28.5] | 23.3 [16.2 to 26.4]
Statistical Analysis 1: Comparison: Control Gefitinib vs Experimental: Gefitinib in Combination With Olaparib; Test type: Superiority; p = 0.3455, Log Rank; Hazard Ratio (HR) = 1.220, 95% CI 2-sided [0.806 to 1.845]

3. Secondary Outcome: Best Global Response During Treatment Period
Description: To evaluate the best global response of the treatment as measured by investigator-assessed overall response rate (ORR) according to RECIST v1.1. Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0) for target lesions and assessed by MRI: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Overall Response (OR) = CR + PR
Time Frame: From the date of randomization until end of follow up, up to 30 months
Measure: Number; unit: participants
Arm/Group | Control Gefitinib | Experimental: Gefitinib in Combination With Olaparib
Number analyzed (Participants) | 91 | 91
participants
  Complete Response | 2 | 1
  Partial Response | 59 | 59
  Stable disease | 21 | 12
  Progressive Disease | 6 | 8
  Not evaluable | 3 | 11

ADVERSE EVENTS:
Time Frame: 37 months
Description: The severity of AE will be determined using CTCAE version 4.0.
Arm/Group | Control Gefitinib | Experimental: Gefitinib in Combination With Olaparib
All-Cause Mortality (participants affected / at risk) | 10/91 | 9/91
Serious Adverse Events (participants affected / at risk) | 39/91 | 22/91
Other Adverse Events (participants affected / at risk) | 88/91 | 90/91
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Control Gefitinib (N=91) | Experimental: Gefitinib in Combination With Olaparib (N=91)
Hypertension (Vascular disorders) | 2 (2) | 1 (1)
Pericardial effusion (Cardiac disorders) | 1 (1) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Other - Respiratory, Thoracic And Mediastinal Disorders (Respiratory, thoracic and mediastinal disorders) | 10 (10) | 11 (11)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2)
Anemia (Blood and lymphatic system disorders) | 10 (10) | 16 (16)
Bone marrow aplastic (Blood and lymphatic system disorders) | 1 (1) | 1 (1)
Cerebral infart subjects affected (Nervous system disorders) | 1 (1) | 1 (1)
Edema Limbs (General disorders) | 1 (1) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 2 (2) | 3 (3)
Mucositis oral (Gastrointestinal disorders) | 1 (1) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1) | 1 (1)
Gastrointestinal infection (Gastrointestinal disorders) | 1 (1) | 1 (1)
Renal insuficiency (Renal and urinary disorders) | 1 (1) | 1 (1)
Rash acneiform (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 3 (3)
Asthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Control Gefitinib (N=91) | Experimental: Gefitinib in Combination With Olaparib (N=91)
Alanine aminotransferase increased (Investigations) | 28 (28) | 14 (14)
GGT increase (Investigations) | 18 (18) | 15 (15)
Alkaline Phosphatase Increased (Investigations) | 16 (16) | 16 (16)
Aspartate aminotransferase increased (Investigations) | 20 (20) | 10 (10)
Lipasa increased (Investigations) | 7 (7) | 4 (4)
Cough (Respiratory, thoracic and mediastinal disorders) | 37 (37) | 29 (29)
Flu like symptoms (Respiratory, thoracic and mediastinal disorders) | 14 (14) | 5 (5)
Bronchial infection (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 0 (0)
Dysgeusia (Nervous system disorders) | 6 (6) | 14 (14)
Fatigue (General disorders) | 50 (50) | 46 (46)
Fever (General disorders) | 11 (11) | 6 (6)
Nausea (Gastrointestinal disorders) | 23 (23) | 51 (51)
Vomiting (Gastrointestinal disorders) | 17 (17) | 34 (34)
Urinary tract infection (Renal and urinary disorders) | 14 (14) | 11 (11)
Dry skin (Skin and subcutaneous tissue disorders) | 21 (21) | 18 (18)
Alopecia (Skin and subcutaneous tissue disorders) | 12 (12) | 12 (12)
Pruritus (Skin and subcutaneous tissue disorders) | 11 (11) | 13 (13)
Anorexia (General disorders) | 25 (25) | 40 (40)
Paronychia (Infections and infestations) | 15 (15) | 7 (7)
Upper respiratory tract infection (Respiratory, thoracic and mediastinal disorders) | 10 (10) | 4 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No